CLINICAL TRIAL: NCT01565824
Title: Web-based Support During Pregnancy and Early Motherhood in Women With Type 1 Diabetes (MODIAB-web)
Acronym: MODIAB-web
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Diabetes Association (Unknown); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MODIAB-web
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Type 1; Pregnancy; Early Motherhood
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-based support (Experimental): The subjects will get access to a website where they can store blood glucose levels, read specialized information concerning pregnancy and early motherhood, and access a discussion forum for peer support.
  Interventions: Other: web-based support
- Usual care (No Intervention)

INTERVENTIONS:
Other: web-based support
  Arms: Web-based support

SUMMARY:
The aim is to investigate whether the implementation of a web-based support to women with type 1 diabetes during pregnancy and early motherhood can improve well-being and self management of diabetes. Type 1 diabetes is associated with increased medical risks and increased psychosocial pressure in relation to childbearing. There is need for extended support from both health care professionals and peers. Web-based interventions can improve personal capacity and self-management in people with long- term illnesses but are not evaluated in childbearing women with type 1 diabetes. A web site prototype for full-size browsers and mobile devices has been developed through a participatory design by multidisciplinary researchers, health care professionals, experienced mothers with type 1 diabetes and web designers. In a randomised control study the developed web site offering information, communication with health care professionals, person-centred self-care diaries and online social community of included women, is provided to the intervention group in early pregnancy at admission to specialised antenatal clinics at six hospitals in Sweden. A control group will receive standard care (usual care). Total n = 160. Primary outcomes are Well-Being Questionnaire and Diabetes Empowerment Scale. The intervention offers proactive solutions for strengthening patients' decision making of diabetes in daily life during pregnancy and early motherhood, and is expected to increase their wellbeing, personal capacity and knowledge of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* women with type 12 diabetes, included in early pregnancy (first trimester)

Exclusion Criteria:

* women who are illiterate, or do not read and speak Swedish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Diabetes Empowerment Scale (SWE-DES-10) | at inclusion, 7 months after inclusion, 10 months after inclusion, 14 months after inclusion
Well-Being Questionnaire (W-BQ12) | at inclusion, 7 months after inclusion, 10 months after inclusion, 14 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Academy, Institute of Health Care Sciences, Gothenburg, Sweden

REFERENCES:
- [Derived] Adolfsson A, Linden K, Sparud-Lundin C, Larsson PG, Berg M. A web-based support for pregnant women and new mothers with type 1 diabetes mellitus in Sweden (MODIAB-Web): study protocol for a randomized controlled trial. Trials. 2014 Dec 29;15:513. doi: 10.1186/1745-6215-15-513. PMID 25543854